CLINICAL TRIAL: NCT07097831
Title: An Open-label, Single-arm, Fixed-sequence, Single-center Phase I Clinical Trial of HRS-1301 on the Pharmacokinetics of Rosuvastatin Calcium Tablets in Healthy Subjects
Brief Title: A Clinical Trial of HRS-1301 on the Pharmacokinetics of Rosuvastatin Calcium Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1301-102
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: HRS-1301 Tablets; Drug: Rosuvastatin Calcium Tablets

INTERVENTIONS:
Drug: HRS-1301 Tablets — HRS-1301 tablets.
Drug: Rosuvastatin Calcium Tablets — Rosuvastatin calcium tablets.

SUMMARY:
The study was designed to evaluate the pharmacokinetic effects of rosuvastatin calcium tablets after oral administration of HRS-1301 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18-55 years (inclusive).
2. At screening, 18.0 ≤ BMI ≤ 30 kg/m2 (inclusive), and body weight ≥ 50.0 kg and <90.0 kg for males and ≥ 45.0 kg and < 90.0 kg for females.
3. Physical examination, vital signs, electrocardiogram, chest X-ray /CT, abdominal ultrasound, laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function, thyroid function) were normal or abnormal but of no clinical significance.
4. The female subjects were not pregnant or lactating, and the results of pregnancy tests before the test were negative. Those who did not have unprotected sex within two weeks before screening; Female subjects of childbearing potential and men whose partners were women of childbearing age agreed to comply with relevant contraceptive requirements and had no sperm/egg donation plans.
5. Participants were able to communicate well with the investigators, understand and comply with the requirements of the study, and sign the informed consent form.

Exclusion Criteria:

1. Previous medical history or current clinical diagnosis of cardiac, respiratory, endocrine, metabolic, cutaneous, infectious, malignant tumor, hematologic, neurological or psychiatric disorders, metabolic/functional disorders or other diseases.
2. Gastrointestinal, hepatic, or renal disease, as judged by the investigator, or other conditions known to affect the absorption, distribution, metabolism, and excretion of the drug or to impair adherence.
3. Patients with major trauma or surgery within 3 months before screening or planning to undergo surgery during the trial.
4. Patients with specific allergic history (asthma, urticaria, eczema, etc.), or allergic constitution (such as allergic to any drug, food), or known allergic to any ingredient in the study drug.
5. Participants who had used any drugs (including prescription drugs, over-the-counter drugs, herbal medicines, dietary supplements, etc., except regular vitamins and occasional acetaminophen) within 2 weeks before screening, or within 5 half-life periods of the drugs (whichever was longer).
6. Enrolled in a clinical trial of any drug or medical device within 3 months before screening or within 5 half-lives of the drug before screening, whichever is longer.
7. Individuals who have donated ≥ 400 mL blood within 4 weeks before screening, have severe blood loss (blood loss ≥ 400 mL), or have received blood transfusion within 8 weeks before screening.
8. Persons who are scheduled to receive live (attenuated) vaccine within 4 weeks before screening or during the course of the trial.
9. Hepatitis B virus surface antigen, hepatitis C virus IgG antibody, anti-treponema pallidum antibody, human immunodeficiency virus antibody and antigen p24 positive during the screening period.
10. Those with positive alcohol breath test and/or drug abuse screening test at baseline.
11. A history of drug or substance abuse.
12. Potential difficulty in blood collection, with a history of syncope.
13. Investigators, research assistants, pharmacists, research coordinators, or others directly involved in the implementation of the protocol.
14. Any factors considered by the investigator to be unsuitable for participation in the trial.
15. Subjects voluntarily withdraw from the trial due to their own reasons.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time 0 to time t (AUC0-t) | 0 to anticipated 15 days.
Area under the curve from time 0 to time infinity (AUC0-∞) | 0 to anticipated 15 days.
Maximum concentration (Cmax) | 0 to anticipated 15 days.

SECONDARY OUTCOMES:
Time to reach maximum concentration (Tmax) | 0 to anticipated 15 days.
Half-life (t1/2) | 0 to anticipated 15 days.
Apparent clearance (CL/F) | 0 to anticipated 15 days.
Adverse events (AEs) | Baseline up to 19 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided